CLINICAL TRIAL: NCT01443650
Title: A Randomized Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics After Different Single-Dose Subcutaneous Treatments of SAR236553/REGN727 in Healthy Subjects
Brief Title: Injection Site Tolerability, Safety, Pharmacokinetics, Pharmacodynamics in Different Single-Dose Treatments of Alirocumab SAR236553 (REGN727) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKD12275; U1111-1120-0670 (Other: UTN)
Record Dates: First submitted 2011-09-21; First posted 2011-09-30 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2012-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- alirocumab SAR236553 (REGN727) (Formulation A x 1) (Experimental): A single subcutaneous injection of Formulation A
  Interventions: Drug: alirocumab SAR236553 (REGN727)
- alirocumab SAR236553 (REGN727) (Formulation B x 1) (Experimental): A single subcutaneous injection of Formulation B
  Interventions: Drug: alirocumab SAR236553 (REGN727)
- alirocumab SAR236553 (REGN727) (Formulation A x 2) (Experimental): 2 single subcutaneous injections of Formulation A
  Interventions: Drug: alirocumab SAR236553 (REGN727)

INTERVENTIONS:
Drug: alirocumab SAR236553 (REGN727) — Pharmaceutical form:solution Route of administration: subcutaneous

SUMMARY:
Primary Objective:

Injection Site Tolerability

Secondary Objectives:

* To assess the safety profile of alirocumab SAR236553 (REGN727)
* To assess the pharmacokinetic-pharmacodynamic relationship of alirocumab SAR236553 (REGN727)

DETAILED DESCRIPTION:
Total duration for each subject (not including screening) will be approximately 85 days.

ELIGIBILITY:
Inclusion criteria:

* Serum LDL-C levels >100 mg/dL.

Exclusion criteria:

* Subjects indicated for the use of statins according to criteria in Adult Treatment Program (ATP) III Guidelines, as updated in 2004.
* Initiation of a new diet or major change to a previous diet within 4 weeks prior to Screening. Subjects must be willing to maintain a consistent diet for the duration of the study.
* Use of a medication or nutraceutical in order to alter serum lipids within 4 weeks prior to screening, including but not limited to statins, cholesterol absorption inhibitors, fibrates, niacin, bile acid resins, or red yeast rice.
* Fasting serum triglycerides >200 mg/dL measured after an 8-12 hour fast.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pain using Present Pain Intensity (PPI) verbal questionnaire and Visual Analog Scale (VAS) | 15 days
Erythema at injection site by measuring diameter and qualitative assessment | 15 days
Edema at injection site by measuring diameter and qualitative assessment | 15 days

SECONDARY OUTCOMES:
Assessment of PK parameter - time to maximum concentration (tmax) | Up to 85 days
Pharmacodynamics: Change in LDL-C from baseline | Up to 85 days
Number of participants with Adverse Events | Up to 85 days
Assessment of PK parameter - maximum concentration (Cmax) | Up to 85 days
Assessment of PK parameter - area under curve (AUC) | Up to 85 days
Assessment of PK parameter - area under curve versus time curve (AUC0-D29) | Zero to Day 29
Assessment of PK parameter - plasma concentration on Day 29 (C D29) | Day 29
Assessment of PK parameter - terminal elimination half-life (t1/2z) | Up to 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States